CLINICAL TRIAL: NCT03187548
Title: Evaluation of the Demineralizing Effect on Enamel Surface During Orthodontic Treatment With and Without the Addition of Casein Phosphopeptides-Amorphous Calcium Phosphate (CPP-ACP) on: A Randomized Clinical Trial, Split Mouth Design
Brief Title: Evaluation of CPP-ACP Prophylactic Effect on Enamel Surface During Orthodontic Treatment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Abd El-Monem Nasr, Doctor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CPP-ACP_whitespots
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: White Spot Lesion; Enamel Hypomineralization
Keywords: WSL; CPP-ACP
MeSH Terms: conditions — Dental Enamel Hypomineralization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CPP-ACP (Experimental): Casein phosphopeptide amorphous calcium phosphate dental paste
  Interventions: Drug: Casein Phosphopeptide-Amorphous Calcium Phosphate Dental Paste

INTERVENTIONS:
Drug: Casein Phosphopeptide-Amorphous Calcium Phosphate Dental Paste — Application of CPP-ACP on one premolar once every 2 weeks for 3 months.

SUMMARY:
This study is aiming in preventing the formation of WSL associated with orthodontic treatment which occurs to more than 50% of orthodontically treated patients through applying CPP-ACP on the enamel surface once every 2 weeks for 3 months.

DETAILED DESCRIPTION:
CPP-ACP will be applied on premolars to be extracted in orthodontic patients whose treatment plan indicates extraction of at least 2 premolaes of the maxillary arch. Application will continue on one premolar either the right or left one once every 2 weeks for the first 3 months of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* severe crowding
* Increased overjet
* Protruded maxillary base
* Sound maxillary premolars
* medically free
* molar classification class II
* Canine classification class II

Exclusion Criteria:

* spacing of teeth
* Decreased overjet
* Molar classification III Medically compromised patients
* pregnant females
* carious premolars
* hypoplasia

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Effect on enamel surface color | 3 months
  Assessment of the effect of CPP-ACP on enamel surface using ICDAS-II
Effect on enamel surface | 3 mnths
  Assessment of the effect of CPP-ACP on enamel surface using visual analogue scale through digital photograph

SECONDARY OUTCOMES:
Surface texture | 3 months
  Assessment of the effect of CPP-ACP on enamel surface texture using scanning electron microscope
Microhardnes | 3 months
  Assessment of the effect of CPP-ACP on enamel microhardness using Vickers hardness test

CONTACTS AND LOCATIONS:
Overall Officials: Maha Swelam, Bachelor, Principal Investigator — Department of orthodontics

IPD SHARING:
Plan to Share IPD: No